CLINICAL TRIAL: NCT03727815
Title: Mindfulness Meditation to Improve Patient Satisfaction and Post-operative Outcomes in Rhinoplasty Patients: A Randomized Controlled Trial
Brief Title: Effects of Mindfulness Meditation on Rhinoplasty Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired IRB application
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00184434
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Nose Deformity
Keywords: mindfulness; meditation; patient satisfaction; rhinoplasty; pain control; quality of life
MeSH Terms: conditions — Patient Satisfaction; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Pain Management Arm (Experimental): Mindfulness meditation intervention - pain management module: patients will be asked to complete a guided mindfulness meditation phone application intervention that was designed to target pain management through mindfulness.
  Interventions: Other: Mindfulness Pain Management Arm
- Mindfulness Self Esteem Arm (Experimental): Mindfulness meditation intervention - pain management module: patients will be asked to complete a guided mindfulness meditation phone application intervention that was designed to target self esteem through mindfulness.
  Interventions: Other: Mindfulness Self Esteem Arm
- Non-intervention Arm (No Intervention): Patients assigned to the non-intervention arm will not be instructed to use a mindfulness meditation phone application and instead will listen to educational materials.

INTERVENTIONS:
Other: Mindfulness Pain Management Arm — Mindfulness Pain Management intervention: patients will be asked to complete a guided mindfulness meditation intervention using a phone application for 2 weeks prior to participant's scheduled procedure and continue with the pain management mindfulness module for 4 weeks postoperatively with periodic survey assessments using validated psychometric tools.
  Arms: Mindfulness Pain Management Arm
Other: Mindfulness Self Esteem Arm — Mindfulness Self Esteem intervention: patients will be asked to complete a guided mindfulness meditation intervention using a phone application for 2 weeks prior to participant's scheduled procedure and continue with the self esteem mindfulness module for 4 weeks postoperatively with periodic survey assessments using validated psychometric tools.
  Arms: Mindfulness Self Esteem Arm

SUMMARY:
A key factor in determining success of facial plastic plastic surgery is overall patient satisfaction. While a number of patient-reported outcomes tools has been developed, there is still limited research in how physicians can improve patient satisfaction and post-operative outcomes.

The goal of this study is to investigate the effect of a mindfulness meditation phone application on rhinoplasty outcomes. This study will also explore whether mindfulness meditation is a feasible adjunct to current pharmacological modalities of postoperative pain control as well as its potential impact on patient satisfaction. These questions will be answered using a randomized controlled trial.

DETAILED DESCRIPTION:
The field of facial plastic surgery continues to grow as evidenced by the increasing number of services sought by both men and women each year. Among these procedures, rhinoplasty remains one of the most popular surgeries, ranking in the top three most performed cosmetic surgical procedures according to the 2017 Plastic Surgery Statistics Report. A key factor in determining the success of rhinoplasty is overall patient satisfaction. Although many patient-reported outcomes tools have been developed in this space, there is a paucity of research aimed at understanding how physicians can improve patient satisfaction in this patient population. Moreover, strategies to address the psychologic and coping ability for patients undergoing facial plastic surgery have not been investigated. To better provide patient-centered care, physicians should seek to understand the psychosocial impact of perceived nasal deformity and identify patients who may benefit from additional support interventions to complement current rhinoplasty treatment plans.

This is a prospective repeated measures study examining psychosocial status as measured by validated psychometric instruments. The intervention group will participate in mindfulness meditation using a phone application. Assessment of social functioning and quality of life will be conducted using survey instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients who will undergo rhinoplasty
* Patients with access to a smart-phone

Exclusion Criteria:

* Patients younger than 18 years of age
* Non-English speakers
* Patients without smart-phone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Satisfaction with patient's Nose as measured by the FACE-Q Satisfaction with Nose Scale | Baseline (prior to intervention), postoperatively at 2 weeks and 4 weeks
  FACE-Q Satisfaction with Nose scale is a 10-item questionnaire with minimum score 10, maximum score 40 assessing patient satisfaction with patient's nose; each item on the questionnaire can be answered between a range of 1 (very dissatisfied) to 4 (very satisfied) with higher scores indicating greater satisfaction with patient's nose
Change in Patient Satisfaction with patient's Nose as measured by the Rhinoplasty Outcome Evaluation scale | Baseline (prior to intervention), postoperatively at 2 weeks and 4 weeks
  Rhinoplasty Outcome Evaluation scale is a 6-item questionnaire with minimum score of 0 and maximum score of 24 assessing patient satisfaction with patient's nose; each item on the questionnaire can be answered between a range of 0 to 4 regarding statements related to patient's nose with higher scores indicating greater satisfaction with patient's nose

SECONDARY OUTCOMES:
Pain as measured by Visual Analog Scale | Postoperatively at day 2, 2 weeks and 4 weeks
  Pain Visual Analog Scale - single-item question ranging from 0 to 100 with greater numbers indicating more pain experienced after surgery
Pain Control as measured by Prescription Analgesic Use | Single measure postoperatively at routine follow-up appointment up to 1 month post procedure
  Pain control as measured by prescription analgesic use will be confirmed at the routine postoperative follow-up appointment by prescription pain medication pill-counting to ascertain analgesic usage over the recovery period
Screen for Body Dysmorphic Disorder as measured by the Body Dysmorphic Disorder Questionnaire | Baseline (prior to intervention)
  Body Dysmorphic Disorder Questionnaire (BDDQ) - 4-item questionnaire with yes/no responses related to concerns about physical appearance; a "positive" screen per the BDDQ instruction manual suggests the possibility of body dysmorphic disorder but is not diagnostic
Change in Anxiety as measured by the State-Trait Anxiety Inventory | Baseline (prior to intervention), 2 weeks, 4 weeks
  State-Trait Anxiety Inventory - 20-item questionnaire with minimum score of 20 and maximum score of 80 (with higher scores meaning more anxiety) intended to measure state anxiety with categorical responses ranging from "never" to "very much so" (4-point Likert scale) in regards to statements about how one feels at the current moment (state) and more generally (trait)
Change in Mindfulness as measured by the Cognitive and Affective Mindfulness Scale-Revised | Baseline (prior to intervention), 2 weeks, 4 weeks
  Cognitive and Affective Mindfulness Scale-Revised - 12-item questionnaire with a minimum score of 12 points and a maximum score of 48 tallied by categorical responses ranging from "rarely/not at all" (1) to "almost always" (4) per item regarding statements about one's experience of mindfulness where higher scores indicate greater mindful qualities
Early Postoperative Symptoms as measured by FACE-Q Recovery Early Symptoms Scale | Postoperatively at day 2
  FACE-Q Recovery Early Symptoms scale - 17-item questionnaire with minimum score 17 and maximum score 68 assessing early symptoms after surgery; each item on the questionnaire can be answered between a range of 1 (not at all) to 4 (extremely) regarding specific symptoms participants may or may not be experiencing after surgery with higher scores indicating greater discomfort, more symptoms, or both
Patient Satisfaction with Doctor as measured by FACE-Q Satisfaction with Doctor Scale | Postoperatively at 4 weeks
  FACE-Q Satisfaction with Doctor scale - 10-item questionnaire with minimum score 10 and maximum score 40 assessing patient satisfaction with patient's doctor; each item on the questionnaire can be answered between a range of 1 (definitely disagree) to 4 (definitely agree) with higher scores indicating greater satisfaction with patient's doctor

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ishii, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins - Green Spring Station, Lutherville-Timonium, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosmetic Surgery National Data Bank Statistics. Aesthet Surg J. 2016 Apr;36 Suppl 1(Suppl 1):1-29. doi: 10.1093/asj/36.Supplement_1.1. No abstract available. PMID 27069249
- [Background] Klassen AF, Cano SJ, Scott A, Snell L, Pusic AL. Measuring patient-reported outcomes in facial aesthetic patients: development of the FACE-Q. Facial Plast Surg. 2010 Aug;26(4):303-9. doi: 10.1055/s-0030-1262313. Epub 2010 Jul 27. PMID 20665408
- [Background] Perry F, Parker RK, White PF, Clifford PA. Role of psychological factors in postoperative pain control and recovery with patient-controlled analgesia. Clin J Pain. 1994 Mar;10(1):57-63; discussion 82-5. doi: 10.1097/00002508-199403000-00008. PMID 8193445
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896
- [Background] Guendelman S, Medeiros S, Rampes H. Mindfulness and Emotion Regulation: Insights from Neurobiological, Psychological, and Clinical Studies. Front Psychol. 2017 Mar 6;8:220. doi: 10.3389/fpsyg.2017.00220. eCollection 2017. PMID 28321194
- [Background] Zeidan F, Vago DR. Mindfulness meditation-based pain relief: a mechanistic account. Ann N Y Acad Sci. 2016 Jun;1373(1):114-27. doi: 10.1111/nyas.13153. PMID 27398643